CLINICAL TRIAL: NCT03987217
Title: Creatine Supplementation With Resistance Training: A Novel Approach to Improving Body Composition and Associated Health Outcomes Among Prostate Cancer Patients
Brief Title: Resistance Training +/- Creatine for Metastatic Prostate Cancer Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCI120424; NCI-2019-02877 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HCI120424 (Other: Huntsman Cancer Institute/University of Utah); P30CA042014 (NIH)
Record Dates: First submitted 2019-06-03; First posted 2019-06-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Fatigue; Metastatic Prostate Carcinoma; Sedentary Lifestyle; Stage IV Prostate Cancer AJCC (American Joint Committee on Cancer) v8; Stage IVA Prostate Cancer AJCC (American Joint Committee on Cancer) v8; Stage IVB Prostate Cancer AJCC (American Joint Committee on Cancer) v8
MeSH Terms: conditions — Fatigue; Prostatic Neoplasms; Sedentary Behavior | interventions — Creatine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (resistance training) (Experimental): Patients complete POWER resistance training program sessions twice weekly over 30-60 minute each for 12 weeks.
  Interventions: Behavioral: Exercise Intervention; Other: Questionnaire Administration
- Group II (resistance training, creatine supplementation) (Experimental): Patients complete POWER resistance training program sessions twice weekly over 30-60 minutes each for 12 weeks and receive creatine monohydrate supplementation given orally 4 times daily during week 1, and then QD (once per day) during weeks 2-12.
  Interventions: Dietary Supplement: Creatine Monohydrate; Behavioral: Exercise Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Dietary Supplement: Creatine Monohydrate — Given orally
  Other Names: Creatine Supplement
  Arms: Group II (resistance training, creatine supplementation)
Behavioral: Exercise Intervention — Complete POWER resistance training program
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well resistance training with or without creatine monohydrate supplement works in improving body composition and health outcomes in patients with prostate cancer that has spread to other places in the body. Resistance training, with or without creatine monohydrate supplement, may help to improve feelings of tiredness and overall physical function in patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the change in lean mass with 12 weeks of creatine supplementation + resistance training compared to resistance training alone.

SECONDARY OBJECTIVES:

I. To evaluate change in other body composition variables (i.e. fat mass, fat-free mass, percent body fat, appendicular lean mass) with 12 weeks of creatine supplementation + resistance training compared to resistance training alone.

II. To evaluate the change in health outcomes associated with body composition (i.e. physical function, fatigue, insulin regulation) with 12 weeks of creatine supplementation + resistance training compared to resistance training alone.

III. To examine associations between creatine supplementation use and changes in biomarkers linked with prostate cancer progression (prostate specific antigen [PSA] and markers of the immune system and allostatic load).

IV. To evaluate the degree of adherence to the creatine supplementation protocol.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients complete Personal Optimism with Exercise Recovery (POWER) resistance training program sessions twice weekly over 30-60 minute each for 12 weeks.

GROUP II: Patients complete POWER resistance training program sessions twice weekly over 30-60 minutes each for 12 weeks and receive creatine monohydrate supplementation orally (PO) 4 times daily during week 1, and then once daily (QD) during weeks 2-12.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic prostate cancer patients who have not met criteria for disease progression on ongoing systemic therapy.
* Currently treated with CYP17A1 inhibitors, surgical castration or medical castration with GnRH (gonadotropin-releasing hormone) agonists/antagonists, or androgen receptor blockers. Must have started the current regimen at least 12 weeks prior to enrollment.
* Confirmation by the patient's treating oncologist that the patient is able to start the exercise program.
* Regular access to an electronic device with internet service and ability for video calls (i.e. computer, smart phone, ipad, tablet, etc).
* Access to an active MyChart account or the willingness to create an account for the purposes of the trial.
* Must be able to read and understand English.
* Willingness to engage in a home-based resistance exercise program two days per week.
* If randomized to the creatine + resistance training group, willingness to take creatine monohydrate supplementation for the duration of the 12 week trial and avoid taking additional creatine-containing supplementation or other supplementation during the study period.
* If randomized to the resistance training group without creatine supplementation, willingness to avoid taking creatine monohydrate supplementation or additional creatine-containing supplementation or other supplementation during the study period.
* For participants randomized to the creatine arm willingness to complete and submit Weekly Creatine Supplementation logs to study personnel via email, fax, or in person.
* Willingness to complete two assessment sessions (baseline and end-of-study).
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Treatment with cytotoxic chemotherapy within 12 weeks prior to enrollment.
* Estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73 m^2.
* Metastatic disease that, in the opinion of the treating oncologist, may obstruct compliant participation in the exercise program (i.e. extensive bone disease).
* Current or planned treatment with radiation therapy. *Subjects who may later require radiation therapy for their health and wellbeing during the course of the trial may be allowed to continue on trial, pending consultation with the PI, treating oncologist, and medical monitor (and DSMC as applicable).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Change in lean mass | Baseline to 12 weeks post intervention
  Assessed by whole-body dual x-ray absorptiometry (DXA) scan.

SECONDARY OUTCOMES:
Change in fat mass | Baseline to 12 weeks post intervention
  Assess body composition by whole-body DXA (dual x-ray absorptiometry) scan.
Change in fat-free mass | Baseline to 12 weeks post intervention
  Assess body composition by whole-body DXA (dual x-ray absorptiometry) scan.
Change in percent body fat | Baseline to 12 weeks post intervention
  Assess body composition by whole-body DXA (dual x-ray absorptiometry) scan.
Change in appendicular lean mass | Baseline to 12 weeks post intervention
  Assess body composition by whole-body DXA (dual x-ray absorptiometry) scan.
Change in physical function | Baseline to 12 weeks post intervention
  Assessed by physical performance battery testing
Change in fatigue | Baseline to 12 weeks post intervention
  Assessed by Functional Assessment of Chronic Illness Therapy Fatigue (FACIT Fatigue Scale, version 4) questionnaire which is a patient-reported measurement of change in fatigue. Level of fatigue is rated from 0 (not at all) to 4 (very much).
  FACIT-Fatigue Subscale Scoring Guidelines (Version 4)
  1. Record answers in "item response" column. If missing, mark with an X
  2. Perform reversals as indicated, and sum individual items to obtain a score.
  3. Multiply the sum of the item scores by the number of items in the subscale, then divide by the number of items answered. This produces the subscale score.
  4. The higher the score, the better the QOL.
Change in insulin regulation | Baseline to 12 weeks post intervention
  Assessed by Homeostatic Model Assessment of Insulin Resistance assessment.
Change in serum PSA (prostate specific antigen) markers of the immune system and allostatic load | Baseline to 12 weeks post intervention
  Assessed by PSA lab
Plasma markers of allostatic load: Interleukin-6 (IL-6) | Baseline to 12 weeks post intervention
  Change in IL-6 will be assessed by serum IL-6 testing.
Plasma markers of allostatic load: Insulin | Baseline to 12 weeks post intervention
  Changes in insulin will be assessed by serum insulin testing.
Plasma markers of allostatic load: Glucose | Baseline to 12 weeks post intervention
  Changes in glucose will be assessed by serum glucose testing.
Total percent of creatine supplementation consumed at end of study | Baseline up to 12 weeks post intervention
  Assessed by submission of supplementation logs and research pharmacy measurements of remaining creatine in the supplementation containers that will be returned by patients at the end-of-study assessment session. Pharmacy creatine measurements will be documented in Vestigo.
Plasma markers of the immune system | Baseline up to 12 weeks post intervention
  Changes in plasma markers of the immune system.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Coletta, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No